CLINICAL TRIAL: NCT06055062
Title: Cerebral Magnetic Resonance Spectroscopy at Term Corrected Age and Dysexecutive Syndrome in Very Preterm Children at 5.5-years-old: EPIPAGE2 and EPIRMEX Cohort Study
Brief Title: Cerebral Magnetic Resonance Spectroscopy at Term Corrected Age and Dysexecutive Syndrome in Very Preterm Children at 5.5-years-old
Acronym: Spectro5-5
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM22_0508
Record Dates: First submitted 2023-09-20; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Compared to term-born peers, very preterm children generally perform poorly in executive functions, with a significant impact on learning at school and quality of life. These EF deficits are related to microstructural abnormalities in white matter and subcortical brain structure.

Objective: To investigate if an alteration of cerebral metabolism in very premature at term corrected-age correlates to executive dysfunctions at school age.

Design, setting, patients: Very preterm patients eligible for Epirmex underwent cerebral Magnetic Resonance Imaging at term-equivalent age and 1H-MRS using a monovoxel technique. The volumes of interest were the posterior periventricular white matter zone and the basal ganglia and thalamus The ratios of N Acetyl Aspartate (NAA) to Choline (cho), NAA to Creatine(Cre), Cho to Cr, and Lac (Lactate) to Cr were calculated.

Main outcome measures: Survival at 5 ½ years with or without neurodevelopmental disabilities (composed of cerebral palsy, visual, hearing, cognitive deficiency, behavioral difficulties, or developmental coordination disorders) were described. The executive functions were assessed using two indices from the Wechsler Intelligence Scale measured in the EPIPAGE 2 cohort at age five-and one-half years: the Working Memory Index (WMI) and the Fluid Reasoning Index (FRI).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria form EPIPAGE2 and EPIRMEX
* Children who underwent spectroscopy with regions of interest analyzed: periventricular zone, gray nuclei, brainstem.
* Children who received a complete cognitive assessment in EPIRMEX (integrated assessment identical to that planned in EPIPAGE2) at age 5 ½.

Non-inclusion Criteria:

* Children with severe karyotype abnormalities.
* Children with central nervous system malformations diagnosed antenatally or on neonatal tests
* Children with severe cerebral palsy or major neurosensory (blindness, profound deafness...) not allowing children to take the tests scheduled at age 5 ½.

Ages: 66 Months to 66 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A French cohort preterm population from the EPIPAGE-2 study.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
neurodevelopmental development | 1 month
  neurodevelopmental development will be judged on the presence of neurodevelopmental disorders as follows :
  * severe or moderate disorders
  * mild disorders
  * absence of disorders

SECONDARY OUTCOMES:
Explored disabilities | 1 month
  Explored disabilities will be classified as follows :
  * motor disabilities
  * cognitive disabilites
  * sensory disabilities
  * behavioral disorders
Schooling | 1 month
  Schooling will be judged on the following criteria: type of establishment, specific assistance.

IPD SHARING:
Plan to Share IPD: No